CLINICAL TRIAL: NCT00057603
Title: Pilot Study of DBS for Treatment-Refractory OCD
Brief Title: Deep Brain Stimulation for Treatment-Resistant Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH064161 (NIH); R21MH064161 (NIH); DATR A5-ETMA
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Participants receive deep brain stimulation treatment for 30 months.
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Deep brain stimulation sends electrical signals to specific parts of the brain, which block the impulses that cause neurological dysfunction.

SUMMARY:
This study will evaluate the use of Deep Brain Stimulation (DBS) to reduce symptom severity and enhance the quality of life for patients with treatment-resistant obsessive compulsive disorder (OCD).

DETAILED DESCRIPTION:
Despite advances in pharmacological and behavioral therapies for OCD, a substantial number of patients fail to improve significantly following years of conventional and experimental interventions. For some patients, stereotactic neurosurgery is the only promising option available. Although this procedure has relatively few side effects in the majority of OCD patients and may lead to enduring benefits, its effects on brain tissue and function are irreversible. Bilateral deep brain stimulation (DBS) is an adjustable and partially reversible procedure that may be a more effective treatment for patients with OCD. This study will determine the effectiveness, safety, and tolerability of DBS in patients with treatment-refractory OCD.

Participants receive DBS treatment for 30 months. Obsessive Compulsive scales, depression scales, neuropsychological evaluations, and surveys are used to assess participants.

Participants are monitored for 2 years after DBS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Intractable, malignant, and treatment refractory OCD that has caused substantial suffering and a reduction in the patient's psychosocial functioning for > 5 years
* Poor prognosis without neurosurgical intervention
* Failed an adequate trial of clomipramine and at least two of the following selective serotonin reuptake inhibitors (SSRIs): fluoxetine, fluvoxamine, citalopram, sertraline, and paroxetine. Additionally, patients must have failed augmentation treatment with at least one of the above drugs for 1 month with at least two of the following: clonazepam, haloperidol, risperidone, olanzapine, and gabapentin.
* Willingness to undergo augmentation treatment with a low-dose neuroleptic if tics are present prior to surgery
* Failed an adequate trial of cognitive behavioral therapy/exposure response prevention while taking clomipramine and an SSRI

Exclusion Criteria:

* Current or lifetime Axis I diagnosis that substantially complicates function, treatment, or the subject's ability to comply with study procedures, or may lead to serious adverse events such as overdose, attempted suicide, or other potentially threatening behaviors
* Diagnosis and/or treatment for depression within the past year. Patients with a more distant history of depression will not be excluded.
* Previous neurosurgical procedure or AXIS III diagnosis of brain pathology
* Implants that contain electrical circuitry, generate electrical signals, and/or have metal parts
* Nonremovable body jewelry
* Anticoagulants or other medications that would put patients at risk for surgery-related complications
* Diathermy for physical therapy
* Pregnancy

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2001-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Obsessive-compulsive scales, depression scales, neuropsychological evaluations, and survey | Measured pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Ward, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Medicine, Gainesville, Florida, United States

REFERENCES:
- [Derived] Vora AK, Ward H, Foote KD, Goodman WK, Okun MS. Rebound symptoms following battery depletion in the NIH OCD DBS cohort: clinical and reimbursement issues. Brain Stimul. 2012 Oct;5(4):599-604. doi: 10.1016/j.brs.2011.10.004. Epub 2011 Nov 4. PMID 22305344
- [Derived] Goodman WK, Foote KD, Greenberg BD, Ricciuti N, Bauer R, Ward H, Shapira NA, Wu SS, Hill CL, Rasmussen SA, Okun MS. Deep brain stimulation for intractable obsessive compulsive disorder: pilot study using a blinded, staggered-onset design. Biol Psychiatry. 2010 Mar 15;67(6):535-42. doi: 10.1016/j.biopsych.2009.11.028. Epub 2010 Feb 8. PMID 20116047